CLINICAL TRIAL: NCT01768832
Title: Exercise and Parkinson's: Comparing Interventions and Exploring Neural Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01NS077959-01A1 (NIH)
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; walking; fMRI; exercise; dance; treadmill
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise Test; Aryl Hydrocarbon Receptor Nuclear Translocator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treadmill (Experimental): Individuals assigned to the Treadmill group will complete two one hour treadmill training sessions per week for 12 weeks.
  Interventions: Behavioral: Treadmill
- Tango (Experimental): Individuals assigned to the Tango group will complete two one hour dance classes twice per week for 12 weeks.
  Interventions: Behavioral: Tango
- Stretching (Active Comparator): Individuals assigned to Stretching will complete two one hour stretching classes per week for 12 weeks.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Treadmill
  Arms: Treadmill
Behavioral: Tango
  Arms: Tango
Behavioral: Stretching
  Arms: Stretching

SUMMARY:
Parkinson disease (PD) is characterized by substantial disability and reduced quality of life, both of which can be attributed in large part to difficulties with walking. Evidence suggests that exercise may be an important addition to traditional treatments, particularly with respect to addressing walking problems. In particular, dance and treadmill training have been individually shown to improve walking performance and quality of life. At present it is not clear whether dance or treadmill training have similar effects or if one is superior to the other. Furthermore, our understanding of the means by which these exercise interventions convey benefits is extremely limited. This study aims to address these knowledge gaps by directly comparing dance, treadmill training and stretching (control group). The primary area of interest is the effects on gait, with secondary measures of disease severity, balance, and quality of life. The investigators will determine not only the effects of the interventions on walking performance, but will also investigate the effects of the interventions on connections between different parts of the brain and on brain function during imagined walking tasks using functional magnetic resonance imaging (fMRI). Participants will be randomly assigned to dance, treadmill training, or a stretching/flexibility control group. Participants will be assessed over a period of 6 months at 3 different time points. The investigators hypothesize that both dance and treadmill training will lead to improvements in forward walking, but that dance will result in greater improvements in backward walking compared to treadmill training. Furthermore, the investigators hypothesize that the tango and treadmill interventions will have different effects of brain function and brain connections. The investigators expect dance to enhance the activity and connections of particular brain regions and treadmill training to enhance activity and connections of different brain regions. The investigators do not expect changes in brain activity or connections in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of Parkinson disease
2. at least grade 3/5 strength and normal joint ranges of motion in both legs,
3. vision corrected to 20/40 or better,
4. able to walk independently for 10 feet with or without an assistive device, 5) normal gross somatosensory function in the feet (2-point discrimination, vibration, joint kinesthesia, and light touch),

6) no history of vestibular disease, 7) no evidence of dementia

Exclusion Criteria:

1. medical condition for which exercise is contraindicated,
2. evidence of abnormality other than PD-related changes on brain imaging,
3. history or evidence of neurological deficit other than PD that could interfere, such as previous stroke or muscle disease,
4. history or evidence of orthopedic or muscular problem,
5. failed to pass magnetic resonance imaging screening procedure

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gammon M Earhart, PhD, PT, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Rawson KS, McNeely ME, Duncan RP, Pickett KA, Perlmutter JS, Earhart GM. Exercise and Parkinson Disease: Comparing Tango, Treadmill, and Stretching. J Neurol Phys Ther. 2019 Jan;43(1):26-32. doi: 10.1097/NPT.0000000000000245. PMID 30531383
- [Derived] Earhart GM, Duncan RP, Huang JL, Perlmutter JS, Pickett KA. Comparing interventions and exploring neural mechanisms of exercise in Parkinson disease: a study protocol for a randomized controlled trial. BMC Neurol. 2015 Feb 5;15:9. doi: 10.1186/s12883-015-0261-0. PMID 25652002

RESULTS

PARTICIPANT FLOW:
Groups:
- Treadmill: Individuals assigned to the Treadmill group will complete two one hour treadmill training sessions per week for 12 weeks.
  Treadmill
- Tango: Individuals assigned to the Tango group will complete two one hour dance classes twice per week for 12 weeks.
  Tango
- Stretching: Individuals assigned to Stretching will complete two one hour stretching classes per week for 12 weeks.
  Stretching
Period: Overall Study
Arm/Group | Treadmill | Tango | Stretching
Started | 41 | 43 | 35
Completed | 31 | 39 | 26
Not Completed | 10 | 4 | 9

BASELINE CHARACTERISTICS:
Population: We analyzed baseline data only from those participants who completed at least the first 3 months of the 6 months study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treadmill | Tango | Stretching | Total
Number analyzed (Participants) | 31 | 39 | 26 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.52 (9.54) | 66.73 (9.52) | 66.18 (7.30) | 67.16 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 12 | 40
  Male | 17 | 25 | 14 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 30 | 39 | 26 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 29 | 39 | 23 | 91
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Disease Duration [Mean (Standard Deviation); unit: years] — Years since being diagnosed with Parkinson's disease
  years | 5.59 (3.81) | 6.10 (4.82) | 4.40 (5.04) | 5.47 (4.59)

OUTCOME MEASURES:

1. Primary Outcome: Walking Velocity at Baseline and 3 Months
Description: Walking velocity during forward and backward walking as determined by a computerized mat.
Time Frame: 0 and 3 months
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 31 | 39 | 26
cm/sec
  Baseline Forward Walking Velocity | 103.28 (4.67) | 104.53 (3.92) | 111.21 (3.81)
  Forward Walking Velocity at 3 months | 109.57 (4.65) | 103.36 (4.21) | 110.52 (5.02)
  Baseline Backward Walking Velocity | 63.45 (4.22) | 60.80 (3.70) | 65.17 (4.60)
  Backward Walking Velocity at 3 months | 64.89 (3.72) | 71.87 (4.83) | 75.17 (6.69)

2. Secondary Outcome: Blood Oxygen Level Dependent Signal at Baseline to 3 Months
Description: Measure of the ratio of oxygenated to deoxygenated blood in areas of the brain at a specific time. Used as an indirect assessment of brain activity and connections. Higher values indicate more brain activity in the brain areas of interest.
Time Frame: 0 and 3 months
Population: Due to issues with data quality related to head movement while in the MRI scanner, we had a limited numbers of participants in each group with usable MRI data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 11 | 13 | 13
ratio
  Bold Signal at Baseline in Primary Motor Cortex | .110 (.165) | .043 (.255) | .095 (.307)
  Bold Signal at 3 months in Primary Motor Cortex | .126 (.246) | .111 (.242) | .117 (.159)

3. Secondary Outcome: Mini Balance Evaluation Systems Test (Mini-BESTest) at Baseline and 3 Months
Description: The Mini Balance Evaluation Systems Test (Mini-BESTest) is a clinical assessment of balance ability. Score range from 0 to 28 with higher scores indicating better balance.
Time Frame: 0 and 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 31 | 39 | 26
score on a scale
  MiniBEST at baseline | 19 [15.5 to 21.5] | 19 [17 to 21] | 20 [18 to 22]
  MiniBESTest at 3 months | 19 [17 to 23] | 19 [17 to 22.5] | 21 [18.25 to 22.75]

4. Secondary Outcome: PDQ-39 Scores at Baseline and 3 Months
Description: The Parkinson Disease Quality of Life Questionnaire is a 39-item tool rating quality of life with higher scores indicating better quality of life. Scores range from 0 to 195.
Time Frame: 0 and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 31 | 39 | 26
score on a scale
  PDQ-39 at baseline | 19.22 (2.71) | 18.33 (1.89) | 16.30 (1.86)
  PDQ-39 at 3 months | 17.86 (2.41) | 18.80 (1.85) | 16.39 (2.35)

5. Secondary Outcome: Movement Disorder Society Unified Parkinson Disease Rating Scale Subscale III at Baseline to 3 Months
Description: The Movement Disorder Society Unified Parkinson Disease Rating Scale - Subscale III is a standardized rating of motor symptom severity in Parkinson disease. Scores range from 0 to 132 with higher scores being worse, i.e. higher scores indicate more severe disease.
Time Frame: 0 and 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 31 | 39 | 26
score on a scale
  MDS-UPDRS-III at baseline | 37 [30 to 41.5] | 37 [29.5 to 41.5] | 38 [33.25 to 44.5]
  MDS-UPDRS-III at 3 months | 33 [25 to 39] | 33 [27.5 to 41.5] | 33 [27.25 to 38]

6. Secondary Outcome: Mini Balance Evaluation Systems Test (Mini-BESTest) at 3 and 6 Months
Description: as for outcome 3
Time Frame: 3 and 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 29 | 36 | 23
score on a scale
  MiniBESTest at 3 months | 20 [17 to 23] | 20 [17 to 23] | 21 [18.5 to 23]
  MiniBESTest at 6 months | 20 [17 to 22] | 19 [18 to 22] | 20 [18 to 21]

7. Secondary Outcome: Movement Disorder Society Unified Parkinson Disease Rating Scale Subscale III at 3 Months and 6 Months
Description: as for outcome 5
Time Frame: 3 and 6 months
Population: Analysis included only participants who completed the study visit at the six month time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 29 | 36 | 23
score on a scale
  MDS-UPDRS-III at 3 months | 32 [24 to 38] | 32 [27 to 39.25] | 33 [27 to 38.5]
  MDS-UPDRS-III at 6 months | 32 [27 to 40] | 35 [28.75 to 41.25] | 38 [28.5 to 44]

8. Secondary Outcome: PDQ-39 Scores at 3 Months and 6 Months
Description: as for outcome 4
Time Frame: 3 and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 29 | 36 | 23
score on a scale
  PDQ-39 at 3 months | 17.86 (2.41) | 18.80 (1.85) | 16.39 (2.35)
  PDQ-39 at 6 months | 12.66 (2.41) | 19.20 (1.75) | 9.33 (1.40)

9. Secondary Outcome: Walking Velocity at 3 Months and 6 Months
Description: Walking velocity during forward and backward walking as determined by a computerized mat.
Time Frame: 3 and 6 months
Population: Analysis included only those participants who completed the 6 month visit.
Measure: Median (Inter-Quartile Range); unit: cm/sec
Arm/Group | Treadmill | Tango | Stretching
Number analyzed (Participants) | 29 | 36 | 23
cm/sec
  Forward Walking Velocity at 3 months | 116.7 [10.7 to 128.5] | 109.7 [93.73 to 123.5] | 111.6 [101.4 to 125.5]
  Forward Walking Velocity at 6 months | 113.9 [102 to 125.7] | 108.4 [89.33 to 124.9] | 117 [104.6 to 126]
  Backward Walking Velocity at 3 months | 78.8 [60.3 to 95.1] | 67.8 [54.05 to 79.4] | 73.4 [55.05 to 87.95]
  Backward Walking Velocity at 6 months | 74.2 [60.4 to 95.8] | 70.3 [44.93 to 81.43] | 68.2 [55.05 to 89.5]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Arm/Group | Treadmill | Tango | Stretching
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/39 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/39 | 0/26
Other Adverse Events (participants affected / at risk) | 0/31 | 0/39 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT01768832/Prot_SAP_000.pdf